CLINICAL TRIAL: NCT05211778
Title: Post-Operative Patient-Centred Care Education Administration in Head and Neck Cancer Patients - A Digital Platform
Brief Title: Digital Patient Education Platform in Head and Neck Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Eitan Prisman, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H16-01039
Record Dates: First submitted 2022-01-04; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Head and Neck Cancer
Keywords: Education; Patient Satisfaction; Multimedia; Free flap; Head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Patient Satisfaction

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): This group will continue to receive the routine standard of care during their treatment journey.
- Digital Education Group (Experimental): In addition to the standard of care, this group will complete an audiovisual digital education module during their postoperative stay in hospital.
  Interventions: Behavioral: Digital Education Group

INTERVENTIONS:
Behavioral: Digital Education Group — Multimedia education provided to the intervention group via a digital tablet
  Arms: Digital Education Group

SUMMARY:
Head and neck cancer is a disease that has a particular propensity for treatment-related morbidity. It is hypothesized that patients who are more involved in their care in hospital and who are actively provided with more treatment-related education may report increased satisfaction and have improved overall outcomes. The investigators aim to determine whether delivery of patient-centred education in a multimedia format via a digital platform has an impact on overall satisfaction and perceived quality of medical care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 years old or above
* Patients seen in outpatient clinic who are scheduled to undergo reconstructive head and neck surgeries for a confirmed oral or oropharyngeal cancer diagnosis.

Exclusion Criteria:

* Patients who are unable to use a digital tablet
* Patients who do not speak or read English
* Individuals unable to understand the purpose, methods and conduct of this study
* Patients unwilling to provide informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | From date of surgery until the date of discharge. The number of days patients will remain in hospital after surgery can range from 7-14 days.
  Measured via a 5-point Likert scale from a survey collected on discharge day

SECONDARY OUTCOMES:
Perceived quality of medical care | From date of surgery until the date of discharge. The number of days patients will remain in hospital after surgery can range from 7-14 days.
  Measured via a 5-point Likert scale from a survey collected on discharge day

CONTACTS AND LOCATIONS:
Overall Officials: Eitan Prisman, MD, FRCSC, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No